CLINICAL TRIAL: NCT02233283
Title: Effect of Metabolic Variations Upon the Activity of the Neuroendocrine Reproductive Axis in Normal Female Volunteers
Brief Title: Effect of Modifications of Nutritional Intake Upon Reproductive Hormones in Normal Women
Acronym: Polynut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Francois Pralong, Full professor and Head, Service of Endocrinology, Diabetology and Metabolism, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 43/13; 320030_141065 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2014-07-21; First posted 2014-09-08 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Female Reproductive System Disorder
Keywords: LH pulsatility; Insulin sensitivity; Metabolism; hypercaloric feeding
MeSH Terms: conditions — Insulin Resistance | interventions — Constriction; Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hypercaloric diet and basal (Active Comparator): Volunteers fed a hypercaloric diet for one month will be submitted to a fasting period of ten hours duration
  Interventions: Other: Hypercaloric diet; Other: Basal
- Hypercaloric diet and clamp (Experimental): Volunteers fed a hypercaloric diet for one month will be submitted to a hyperinsulinemic and euglycemic clamp of ten hours duration
  Interventions: Other: Clamp; Other: Hypercaloric diet
- Isocaloric diet and basal (Active Comparator): Volunteers fed a isocaloric diet for one month will be submitted to a fasting period of ten hours duration
  Interventions: Other: Basal; Other: Isocaloric diet
- Isocaloric diet and clamp (Experimental): Volunteers fed a isocaloric diet for one month will be submitted to a hyperinsulinemic and euglycemic clamp of ten hours duration
  Interventions: Other: Clamp; Other: Isocaloric diet

INTERVENTIONS:
Other: Clamp — Volunteers will be submitted to hyperinsulinemic, euglycemic clamp studies of 10 hours duration.
  Other Names: Hyperinsulinemic and euglycemic clamp study
  Arms: Hypercaloric diet and clamp; Isocaloric diet and clamp
Other: Hypercaloric diet — Hypercaloric diet will be conducted during one month, and designed to provide 30% excess in calories compared to daily requirements. It will consist in a high fat, high carbohydrates diet.
  Other Names: Overfeeding
  Arms: Hypercaloric diet and basal; Hypercaloric diet and clamp
Other: Basal — Keeping the volunteers in the fasting state overnight and for the entire duration of the experiment (10 hours)
  Other Names: Fasting
  Arms: Hypercaloric diet and basal; Isocaloric diet and basal
Other: Isocaloric diet — Isocaloric diet will conducted for one month, and designed to provide the calculated daily energy needs
  Other Names: Controlled diet
  Arms: Isocaloric diet and basal; Isocaloric diet and clamp

SUMMARY:
Undernutrition has a known and well recognized negative impact on reproductive hormones, and ultimately fertility. In contrast, much less is known regarding the potential effects of overnutrition on the same hormones. Epidemiological data suggest that overnutrition might have a deleterious impact as well on the fertile potential of affected women, but very little is known about the mechanisms implicated. Such knowledge may be of importance, given the increasing prevalence of overweight and obesity worldwide.

DETAILED DESCRIPTION:
In the present study, the investigators will perform a very detailed study of the minute to minute regulation of hormones of the neuroendocrine reproductive axis in normal young female volunteers. These studies will initially be performed at base line during isocaloric diet, where the stimulation of LH secretion by exogenous insulin will be tested during hyperinsulinemic eugylcemic clamp studies.

The same studies will then be repeated after a period of one month of controlled hypercaloric diet, where volunteers will receive an excess of approximately 30% KCal compared to their calculated daily energy expenditure. it is anticipated that such hypercaloric nutrition will induce a significant decrease in normal insulin sensitivity of these volunteers. Thus, the effect of changing whole body insulin sensitivity on the fine regulation of neuroendocrine reproductive hormones will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

normally cycling young (between 18 and 30 yo) female, with a BMI between 20 and 25 kg/m2.

-

Exclusion Criteria:

* Personal history of endocrine dysfunction (any kind)
* Hormonal contraception
* Pregnancy
* Food allergy (any kind)
* Intense physical activity (>4 hrs/week)
* Smoking

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Luteinizing hormone secretion | Every ten minutes for 10 hours
  The pulsatility of LH will be assessed by measuring LH levels in blood sample obtained every ten minutes over the entire study period (12 hours).

SECONDARY OUTCOMES:
Insulin sensitivity | 10 hours
  Insulin sensitivity will be defined as the rate of glucose infusion required to maintain euglycemia during the hyperinsulinemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Francois P Pralong, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Clinical Research Center, University Hospital, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] van Leckwyck M, Kong W, Burton KJ, Amati F, Vionnet N, Pralong FP. Decreasing Insulin Sensitivity in Women Induces Alterations in LH Pulsatility. J Clin Endocrinol Metab. 2016 Aug;101(8):3240-9. doi: 10.1210/jc.2016-1727. Epub 2016 Jun 16. PMID 27309039